CLINICAL TRIAL: NCT04447612
Title: A Multi-centre Phase II Randomized-controlled Study on Addition of Durvalumab (MEDI4736) to Induction Chemotherapy and Concurrent Chemoradiation and Followed by Maintenance Durvalumab for Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Concurrent Chemoradiation and Durvalumab for Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Victor H.F. Lee, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 19-534
Record Dates: First submitted 2020-06-21; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; Immune checkpoint inhibitors; Chemotherapy; Radiation therapy; Locoregionally advanced
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — durvalumab; Cisplatin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Randomized-controlled trial
Masking Description: No masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Durvalumab arm (Experimental): Induction phase: Durvalumab 1500mg via intravenous infusion every 4 weeks, with chemotherapy gemcitabine 1000mg/m2 on day 1 and day 8 and cisplatin 100mg/m2 on day 1 via intravenous infusion every 3 weeks for 3 cycles.
  Concurrent phase: Durvalumab 1500mg via intravenous infusion every 4 weeks for 2 cycles, with cisplatin 100mg/m2 via intravenous infusion every 3 weeks for 3 cycles.
  Maintenance phase: Durvalumab 1500mg daily via intravenous infusion every 4 weeks for 8 cycles.
  Interventions: Drug: Durvalumab; Drug: Cisplatin; Drug: Gemcitabine
- Standard of care arm (Active Comparator): Induction phase: Chemotherapy with gemcitabine 1000mg/m2 on day 1 and day 8 and cisplatin 100mg/m2 on day 1 via intravenous infusion every 3 weeks for 3 cycles.
  Concurrent phase: Cisplatin 100mg/m2 on day 1 of radiation therapy via intravenous infusion every 3 weeks for 3 cycles.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Durvalumab — Intravenous infusion of durvalumab 1500mg every 4 weeks for 13 cycles (1 year), starting 1 week before start of induction chemotherapy
  Other Names: MEDI4736
  Arms: Durvalumab arm
Drug: Cisplatin — Induction phase: cisplatin 100mg/m2 on day 1 via intravenous infusion every 3 weeks for 3 cycles Concurrent phase: cisplatin 100mg/m2 starting on day 1 of radiation therapy via intravenous infusion every 3 weeks for 3 cycles
Drug: Gemcitabine — Induction phase: gemcitabine 1000mg/m2 on day 1 and day 8 via intravenous infusion every 3 weeks for 3 cycles

SUMMARY:
The investigators propose a phase II randomized-controlled study on using durvalumab in combination with induction chemotherapy followed by concurrent chemoradiation and adjuvant durvalumab, compared to induction chemotherapy followed by concurrent chemoradiation for previously untreated locoregionally advanced stage III to IVA NPC. In parallel, the investigators will also perform collateral tumor and serum biomarker studies which will be correlated with the treatment response. The investigators will collect fresh tumour biopsies at pretreatment, then serially after induction chemotherapy and after concurrent chemoradiation to investigate the change in microenvironment of the tumour and the surrounding inflammatory cells before and after durvalumab. In addition, the investigators will also measure the change in number and intensity of PD-L1-positive circulating tumour cells (CTC) before and after durvalumab and evaluate their correlation with treatment response.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) of the undifferentiated histology is endemic in southern China and southeast Asia including Hong Kong, Taiwan, Singapore and Malaysia, with a peak annual incidence of up to 30 per 100,000 persons. According to global cancer registry, NPC ranked 11th most common among all malignancies in China in 2008 with an incidence of 2.8/100,000 person-years in men and 1.9/100,000 person-years in females. It is highly associated with prior infection with Epstein-Barr virus and thus it is a highly immune-related malignancy. Treatment strategy is mainly based on the disease stage according to the American Joint Committee on Cancer (AJCC)/Union for International Cancer Control (UICC) staging system. In general, stage I-II diseases are treated with radiation therapy alone while stage III-IV diseases are treated with concurrent chemoradiation with or without adjunct chemotherapy (induction or adjuvant). Intensive pretreatment workup including blood hematology and biochemistry, dedicated head and neck imaging with computed tomography and magnetic resonance imaging and positron-emission tomography with integrated computed tomography (PET-CT) and plasma Epstein-Barr virus (EBV) deoxyribonucleic acid (DNA) are essential in high-risk locoregionally advanced diseases to confirm non-metastatic diseases, since the treatment protocol and overall prognosis between locoregionally advanced (stage III-IVA) disease differ significantly from metastatic disease.

Despite intensive radical treatment in the contemporary radiotherapy era with concurrent chemoradiation with or without adjunct chemotherapy, between 15% and 30% of these patients with stage III-IVA disease develop metastatic diseases at distant sites. Further systemic chemotherapy following radical concurrent chemoradiation may not bring survival benefits, attributed by the compromised physique following intensive radical concurrent chemoradiation and the prolonged treatment-related toxicities brought by adjuvant chemotherapy. The recent Hong Kong NPC Study Group NPC-0502 study failed to show survival benefit in patients with post-treatment detectable plasma EBV DNA after a further 6 cycles of adjuvant chemotherapy compared to those who just observed after radical concurrent chemoradiation. On the other hand, induction chemotherapy followed by concurrent chemoradiation may be the more preferred regimen due to the perceived efficacy of eradication of tumor micro-metastasis and early shrinkage of primary tumor and bulky neck nodes, which allow a more radical radiotherapy dose and better coverage of both the primary tumor and neck nodes. Very recently, a China multi-centre phase III randomised-controlled trial demonstrated an improvement in recurrence-free survival and overall survival (OS) with induction chemotherapy gemcitabine plus cisplatin followed by concurrent chemoradiation versus concurrent chemoradiation alone. Nevertheless, new treatment strategies must be developed to improve treatment outcomes of these high-risk patients with stage III-IVA disease, which has become the major research focus in the past decade. A recent meta-analysis demonstrated that induction chemotherapy followed by concurrent chemoradiation improved overall survival compared to concurrent chemoradiation in the era of modern radiotherapy with intensity-modulated radiation therapy (IMRT).

Immune checkpoint inhibitors are now comprehensively and extensively tested in combination with radiotherapy (RT) as well (NCT01935921, NCT01860430). It has been recently known that RT increases the expression of the major histocompatibility complex (MHC). In turn, the MHC class-I restricted tumor antigen-specific cells elicited by RT will upregulate interferons in the tumors. This radiation-induced local inflammation and tumor-specific effector T cells will provide an additional mechanism for tumor control by modification of the tumor vasculature. In addition, RT will increase dendritic cell surface antigen presentation to T cells and production of cytokines leading to recruitment and activation of leucocytes from peripheral blood and extravasation to tumor parenchyma. These are part of the mechanisms of abscopal effect, a phenomenon where the tumors at the sites far away from the irradiated sites also regress after localized radiotherapy. Having learnt from the pivotal PACIFIC trial on the use of consolidation therapy with durvalumab (anti-PD-L1 monoclonal antibody) which confirmed the efficacy and safety of combination of chemoradiation and immunotherapy for stage III non-small-cell lung cancer, it is prime time to consider incorporation of immune checkpoint inhibitors into concurrent chemoradiation for other solid tumors like head and neck squamous cell carcinoma and NPC. In concurrent +/- adjuvant setting for locoregionally advanced NPC, there are at least two clinical trials on immune checkpoint inhibitors for locoregionally advanced disease. The first one is a phase II single-arm study using nivolumab in combination with concurrent chemoradiation with or without by adjuvant nivolumab for up to 3 months at different dose schedules (NCT03267498). A phase III multi-center randomized-controlled trial (RCT) in China on the use of a locally-manufactured PD-1 monoclonal antibody (SHR-1210) every 4 weeks for 12 cycles starting at 4-6 weeks after concurrent chemoradiation for stage III-IVA NPC versus no adjuvant therapy is currently under way (NCT03427827). It is highly expected and eagerly awaited that immunotherapy with immune checkpoint inhibitors will bring a new insight on the adjuvant treatment for NPC.

In view of the above with promising synergy between radiation therapy and immune checkpoint inhibitors, the investigators propose a phase II RCT on adding durvalumab in combination with induction chemotherapy followed by concurrent chemoradiation and adjuvant durvalumab for previously untreated locoregionally advanced NPC. In parallel, the investigators will also perform collateral tumor and serum biomarker studies which will be correlated with the treatment response. The investigators will collect fresh tumour biopsies at pretreatment, then serially after induction chemotherapy and after concurrent chemoradiation to investigate the change in microenvironment of the tumour and the surrounding inflammatory cells before and after durvalumab. In addition, the investigators will also measure the change in number and intensity of PD-L1-positive circulating tumour cells before and after durvalumab and evaluate their correlation with treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have pathologically confirmed, previously untreated stage III-IVA nasopharyngeal carcinoma (staged by American Joint Committee on Cancer/Union International for Cancer Control 8th edition staging classification) who plan to receive radical chemoradiation +/- durvalumab.
2. Fresh frozen tumour and archived formalin-fixed paraffin-embedded (FFPE) nasopharyngeal tumour specimens must be available for PD-L1 expression and/other biomarker correlation studies.
3. Age between 18-75 years. (The age limit set at 75 years because a previous Hong Kong study showed that elderly patient >70 years had poor tolerance to radiotherapy and worse survival for their NPC. Please refer to Sze et al. Radical radiotherapy for nasopharyngeal carcinoma in elderly patients: The importance of co-morbidity assessment Oral Oncology 2012;48:162-167.)
4. Eastern Cooperative Oncology Group Performance Status of 0 or 1
5. All eligible patients must be magnetic resonance imaging of T1, T2 and T1-contrast enhanced sequences of the head and neck region and PET-CT scan within 60 days of study entry
6. Modified Charlson Comorbidity Score <2
7. Adult Comorbidity Evaluation (ACE)-27 Index <2
8. Pre-existing peripheral neuropathy ≤1
9. Baseline creatinine clearance >60ml/min, calculated by Cockcroft-Gault Formula or derived by collection of 24-hour urine.

   Males:

   Creatinine Clearance (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

   Females:

   Creatinine Clearance (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
10. Adequate serum hematological function defined as:

    * Absolute neutrophil count ≥1.5 × 109/l
    * Hemoglobin ≥9.0 g/dl
    * Platelet ≥100 × 109/l
11. Adequate serum biochemical functions defined as:

    * Alanine transferase ≤3 × upper limit of normal range (ULT)
    * Aspartate transferase ≤3 × ULT
    * Total bilirubin ≤2 x ULT
    * Albumin ≥2.8 g/dl
12. For women of childbearing potential, a negative serum or urine pregnancy test within 14 days prior to the start of treatment for their NPC. Women will be considered postmenopausal if they are amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
13. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
14. Body Weight >30kg
15. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
16. Must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment or 5 half-lives, whichever is shorter.
2. Has a diagnosis of severe active scleroderma, lupus, other rheumatologic or autoimmune disease within the past 3 months before study recruitment. Patients with a documented history of clinically severe autoimmune disease or a syndrome requiring systemic steroids or immunosuppressive agents will not be allowed on this study. Subjects with vitiligo or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections are not excluded from the study. Subjects with hypothyroidism stable on hormone replacement are not excluded from this study.
3. Has had a prior monoclonal antibody within 4 weeks or 5 half-lives, whichever is shorter, prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
4. Has had prior chemotherapy or targeted small molecule therapy (including sorafenib or other anti-vascular endothelial growth factor inhibitor) within 3 weeks prior to administration of the study drug or who has not recovered (i.e., ≤Grade 1 or at baseline) from adverse events due to a previously administered agent. *Note: Subjects with permanent ≤Grade 2 toxicities (e.g. neuropathy) or toxicities corrected through routine medical management (e.g. thyroid replacement for hypothyroidism), are an exception to this criterion and may qualify for the study. *Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy. *Note: Subjects with ≤Grade 2 amylase or lipase elevations abnormalities that have no corresponding clinical manifestations (e.g. manifestation of pancreatitis), are an exception to this criterion and may qualify for the study.
5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, indolent lymphomas, or in situ cervical cancer that has undergone potentially curative therapy
6. Has known carcinomatous meningitis (also known as leptomeningeal carcinomatosis).
7. Has an active infection requiring intravenous systemic therapy or hospital admission.
8. Has a history or current evidence of any condition, therapy, or laboratory abnormality, including psychiatric or substance abuse disorder, that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
9. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 31 weeks after the last dose of trial treatment.
10. Has a known history of Human Immunodeficiency Virus (HIV) (HIV type 1/2 antibodies). Routine checking for Anti-HIV type 1 or Anti-HIV type 2 is not mandatory.
11. Untreated hepatitis B infection. Patients with chronic hepatitis B infection (defined as HBsAg positive) are eligible if they have started anti-viral therapy for at least 1 month and is continuing anti-viral treatment throughout the whole duration of this study.
12. Has received a live vaccine 30 days prior to the first dose of trial treatment.
13. Has experienced Grade 4 toxicity on treatment with prior radiation.
14. Has experienced Grade 3-4 intracranial toxicity (hypophysitis or central nervous system toxicity) with either prior intracranial radiation, anti programmed cell death-1 (PD-1), or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibitor therapy.
15. Is taking > 4mg/day of dexamethasone or its equivalent at the start of immunotherapy or has required > 4mg/day of dexamethasone or its equivalent for 3 consecutive days within 1 week of starting treatment.
16. Allergies and adverse drug reaction to the following: History of allergy to study drug components; History of severe hypersensitivity reaction to any monoclonal antibody.
17. Prior systemic therapy utilizing an anti CTLA-4 or PD-1/PD-L1 agent or other forms of immunotherapy.
18. Has had prior radiation therapy
19. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

    1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
    2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician
20. Major surgical procedure (as defined by the Investigator within 28 days prior to the first dose of IP. Local surgery of isolated lesions for palliative intent is acceptable.
21. History of allogenic organ transplantation.
22. History of leptomeningeal carcinomatosis
23. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart).
24. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 36 months
  Progression-free survival

SECONDARY OUTCOMES:
Best objective response | 36 months
  Best objective response
Overall survival | 36 months
  Overall survival
Toxicity profile | 36 months
  Toxicity profile as assessed by Common Terminology Criteria for Adverse Events version 5.0
Changes in the number of PD-L1 positive circulating tumor cells before and after induction chemotherapy and concurrent chemoradiation | 36 months
  Changes in the number of PD-L1 positive circulating tumor cells before and after induction chemotherapy and concurrent chemoradiation

CONTACTS AND LOCATIONS:
Overall Officials: Victor Lee, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.